CLINICAL TRIAL: NCT05464173
Title: Phase Ib/II Study of Chidamide in Combination With Abemaciclib and Endocrinotherapy（Doctor's Choice） in Patients Previously Treated With Palbociclib in HR+/HER2-Relapsed/Metastatic Breast Cancer
Brief Title: Chidamide in Combination With Abemaciclib and Endocrinotherapy（Doctor's Choice） in Breast Cancer Patients Previously Treated With Palbociclib
Acronym: CINDERELLA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biyun Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Biyun Wang, MD, Biyun Wang, MD, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOUNGBC-19
Record Dates: First submitted 2022-06-15; First posted 2022-07-19 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAF (Experimental): endocrinotherapy（doctor's choice） According to the drug insert abemaciclib 150mg or 100mg bid, Chidamide 10-30mg biw.
  Interventions: Drug: Chidamide; Drug: Abemaciclib; Drug: endocrinotherapy（doctor's choice）

INTERVENTIONS:
Drug: Chidamide — 10-30mg biw
Drug: Abemaciclib — 150mg or 100mg bid
Drug: endocrinotherapy（doctor's choice） — According to the drug insert

SUMMARY:
To evaluate the efficacy and safety of chidamide in combination with abemaciclib and endocrinotherapy（doctor's choice） in locally advanced/metastatic HR+/HER2- breast cancer who had failed prior palbociclib therapy

DETAILED DESCRIPTION:
Phase I (Stage Ib). To evaluate the safety and tolerability of chidamide in combination with abemaciclib and endocrinotherapy（doctor's choice） in locally advanced/metastatic HR+/HER2- breast cancer and to determine the recommended phase II dose of this combination regimen.

Stage 2 (Phase II). To determine the efficacy and safety of chidamide in combination with abemaciclib and endocrinotherapy（doctor's choice） in locally advanced/metastatic HR+/HER2- breast cancer with the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants volunteered to participate in this study and signed an informed consent form.
* Female, aged ≥ 18 years.
* ECOG PS score:0-2.
* Expected survival time ≥ 3 months.
* Histologically or cytologically confirmed estrogen receptor positive and/or progesterone receptor positive, HER2-negative loco-regional recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent.
* Prior anti-tumor setting: ① No prior chemotherapy for recurrent or metastatic breast cancer; ② Disease recurrence and/or metastasis during or after palbociclib-based regimen in the (neo)adjutant setting or disease progression during or after palbociclib-based regimen for at least 6 months in the metastatic setting; ③ No more than 3 lines of prior endocrine therapy for recurrent or metastatic breast cancer and meet one of the following requirements: relapse while after the first 2 years of adjuvant endocrine therapy, or disease progression after the first 6 months of latest endocrine therapy for advance or metastatic breast cancer, while on endocrine therapy;
* At least one extracranial measurable lesion defined according to RECIST V1.1 criteria or only bone lesion;
* The functions of vital organs meet the requirements;
* Participants recovered from any AE associated with prior tumor therapy prior to initial administration of the study drug (grade ≤1);

Exclusion Criteria:

* Prior treatment with histone deacetylase inhibitors (HDACi);
* Previously treated with CDK4/6 inhibitors other than palbociclib;
* Leptomeningeal metastasis confirmed by MRI or lumbar puncture;
* Radiographically confirmed central nervous system metastasis; the following conditions were excluded: ① asymptomatic brain metastases not requiring immediate radiotherapy or surgery; ② previously received local therapy (radiotherapy or surgery) for brain metastasis, stable for at least 4 weeks with imaging confirmation without symptomatic treatment (including glucocorticoid, mannitol, bevacizumab, etc.) for more than 2 weeks and clinical symptoms;
* Participants with visceral crises (e.g., lymphangitis carcinoma, bone marrow replacement, leptomeningeal metastasis, diffuse liver metastasis with abnormal liver functions), rapid disease progression, and patients not suitable for endocrine therapy;
* Participants with ascites, pleural effusion and pericardial effusion with clinical symptoms at baseline, requiring drainage within 4 weeks before the first medication;
* Inability to swallow, intestinal obstruction or other factors affecting drug taking and absorption;
* Systematic treatment such as chemotherapy, targeted therapy or other investigational drugs within 4 weeks prior to the start of treatment; endocrine therapy within 2 weeks prior to the start of treatment;
* Participant was diagnosed with any other malignant tumor in the past 5 years prior to the study, except for radically-treated non-melanoma skin cancer, basal cell or squamous cell skin cancer or cervical carcinoma in situ and thyroid papillary carcinoma.
* The participant has undergone major surgical procedures or significant trauma within 4 weeks prior to the start of treatment, or is expected to undergo major surgical treatment;
* Known history of allergy to the drug components of this regimen;
* Infected with active HBV and HCV; participants with stabilized hepatitis B (HBV-DNA lower than 500 IU/mL or copy number <1000 copies/ mL) and cured hepatitis C (negative for HCV RNA) were excluded;
* Have a history of immunodeficiency disease, including HIV positive, or other acquired or congenital immunodeficiency disease, or have a history of organ transplantation;
* Positive baseline pregnancy test; Or participants of reproductive age who were unwilling to use effective contraception during study participation and for at least 3 months after the last dose;
* According to the judgment of the researcher, there are serious concomitant diseases (such as severe hypertension, diabetes, thyroid disease, active infection, etc.) that endanger the patient's safety or affect the patient's completion of the study;
* The researcher determines that the participant is not suitable for the study;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
DLT | 6 weeks
  DLT:dose-limiting toxicity
PFS | 6 weeks
  PFS：progression free survival

SECONDARY OUTCOMES:
ORR | 6 weeks
  Objective response rate (ORR) : Proportion of subjects whose efficacy was evaluated as CR/PR；
DCR | 6 weeks
  Disease control rate (DCR) : Proportion of subjects whose efficacy was assessed as CR/PR/SD；
CBR | 6 weeks
  Clinical benefit rate (CBR) : Proportion of subjects with CR, PR and SD≥24 weeks during the study；
DOR | 6 weeks
  Duration of remission (DoR) : The time from the first assessment of CR or PR to the first assessment of PD or death from any cause；

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No